CLINICAL TRIAL: NCT03247036
Title: Long Survival After Ischemic Stroke and Thombolysis in Catalonia. Differences by Sex
Brief Title: Long-Term Survival After Ischaemic Stroke: Ebrictus Study
Acronym: EBRICTUS
Status: Completed | Type: Observational
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Principal Investigator, Josep Lluís Clua Espuny, PhD Family and Community Medicine, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Other Study IDs: 4R17/017; 17/034 Codi IDIAP: 4R17/017 (Other Grant/Funding Number: SIDIAP 16/9)
Record Dates: First submitted 2017-08-08; First posted 2017-08-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Ischemic Stroke; Thrombolytic (t-PA) Treatment; Gender Bias; Long Term Adverse Effects
MeSH Terms: conditions — Ischemic Stroke; Sexism; Long Term Adverse Effects | interventions — Fibrinolytic Agents; Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: IV thrombolytic (t-PA) treatment vs not — Acute Stroke Protocol
  Other Names: IV thrombolysis; IV thrombolytic (t-PA) treatment

SUMMARY:
A number of large trials have confirmed the benefits of thrombolysis in acute stroke, but there are gender differences. The authors sought to examine the relationship between sex and outcome after thrombolysis.

Previous reports [1-6] concerning sex-related differences in stroke management and outcome are inconsistent and sometimes difficult to interpret, and so the reasons for gender disparities in stroke outcome have remained unclear. Functional outcomes and quality of life after stroke are consistently poorer in women despite adjustment for baseline differences in age and prestroke function, and the fact that comorbidities and clinical outcomes were not different between women and men [3, 7] . Once the reasons for these differences are better understood, intervention might be possible to help provide the best care for all patients. This work is a continuation and extension of the Ebrictus Study [8-10] . Prior work has suggested sex-based differences in thrombolytic therapy in subjects with acute stroke [11] .The authors will explore whether sex might modify the effect of thrombolysis on survival and functional outcomes in patients with acute ischemic stroke [12] beyond the usually evaluated time period of 6 months after stroke and compared this with the group without thrombolytic treatment.

DETAILED DESCRIPTION:
This is a reprospective, observational cohort study including incident strokes from January 1, 2011 to December 31, 2012 and followed up in December 31, 2016. Statistical approaches are used to analyze survival outcomes. It is a longitudinal study of a population-based cohort of all registered cases of a first episode of stroke that occurred in Catalonia (Spain). Demographic Patterns and Epidemic Characteristics. Life expectancy at birth is 81.34 years globally, 78.26 years for men and 84.74 years for women.

Case Definition The definition of stroke corresponds to that set by the World Health Organization.

Patients were included by using the automated operation of the database of patients with a diagnosis code of stroke (I60-I69).

The inclusion criteria were: age ≥ 15 up to ≤ 90; a diagnosis of stroke explicitly recorded in their medical record at any of the registration systems in the health centers; it should be a first stroke episode, and relevant episode information should be available in clinical records: (a) outpatient clinic, (b) hospital clinic, or (c) access to medical/sociosanitary reports.

The variables on which information was collected were grouped as follows: sociodemographic; clinics: type (ischemic or hemorrhagic stroke) and event date (day/month/year); NIHSS score on admission; whether or not there was thrombolytic therapy; duration of hospital stay; hospital discharge destination (home, higher-level acute hospital, long-term care hospital, death and date thereof); pre- and poststroke functional autonomy [the Barthel score was classified as follows: <20 (total dependence), 20-35 (severe dependence), 40-55 (moderate dependence), ≥ 60 (mild dependence), or 100 (independence) registered for preepisode and for discharge in the medical history of the patient, the hospital, or the primary care center]; functional status of the patient at discharge: death, home-autonomous, home address caregiver, referral to another acute hospital, or convalescent center (temporary or long-term stay), and vital status (alive/dead) of the patient, specifying the date (day/month/year) of death, if any.

Statistical Analysis Computerized statistical analysis was undertaken with the following: (1) descriptive basic statistics and standard deviation of key variables stratified by age and sex and (2) differences in functional outcome and its evolution before and after the episode determined the possible effects on mortality and different residual deficits categorized with the statistical Cox regression model. Mortality should be interpreted as overall mortality and cause-specific, no stroke. Patients who died during hospitalization or within the 1st month are considered 'immediate death'. During follow-up the deceased are described as 'subsequent mortality'.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 15 up to ≤ 90;
* usual residence in Catalonia
* and/or assignment to any of the catalonian primary care centers for 5 years at the time of the stroke episode;
* a diagnosis of stroke explicitly recorded in their medical record at any of the registration systems in the health centers of the area; it should be a first stroke episode, and relevant episode information should be available in clinical records: (a) outpatient clinic, (b)hospital clinic, or (c) access to medical/sociosanitary reports.

Exclusion Criteria:

* intracerebral haemorrhage

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients were included by using the automated operation of the database of patients with a diagnosis code of stroke (I60-I69).
Sampling Method: Non-Probability Sample
Enrollment: 21000 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-08-05 (Actual)

PRIMARY OUTCOMES:
Death all causes | January 1, 2011 to December 31, 2016
  Mortality should be interpreted as overall mortality and cause-specific, no stroke. Patients who died during hospitalization or within the 1st month are considered 'immediate death'. During follow-up the deceased are described as 'subsequent mortality'.

CONTACTS AND LOCATIONS:
Locations (1):
- Plan Director Enfermedad Vascular Cerebral, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Dates files

REFERENCES:
- [Background] Clua-Espuny JL, Ripolles-Vicente R, Forcadell-Arenas T, Gil-Guillen VF, Queralt-Tomas ML, Gonzalez-Henares MA, Panisello-Tafalla A, Lopez-Pablo C, Lucas-Noll J; Ebrictus Group. Sex Differences in Long-Term Survival after a First Stroke with Intravenous Thrombolysis: Ebrictus Study. Cerebrovasc Dis Extra. 2015 Oct 9;5(3):95-102. doi: 10.1159/000440734. eCollection 2015 Sep-Dec. PMID 26648964
- [Background] Clua-Espuny JL, Ripolles-Vicente R, Lopez-Pablo C, Panisello-Tafalla A, Lucas-Noll J, Calduch-Noll C, Gonzalez-Henares MA, Queralt-Tomas ML. [Differences in the survival after an episode of stroke treated with thrombolytic therapy. Study Ebrictus]. Aten Primaria. 2015 Feb;47(2):108-16. doi: 10.1016/j.aprim.2014.04.008. Epub 2014 Jun 19. Spanish. PMID 24953174
- [Background] Gonzalez-Henares A, Clua-Espuny JL, Gil-Guillen VF, Panisello-Tafalla A, Queralt-Tomas ML, Ripolles-Vicente R, Lopez-Pablo C, Lucas-Noll J, Equipo de Investigacion Ebrictus Ede I. [Incidence and preventability of haemorrhagic strokes. Results of the Ebrictus register]. Rev Neurol. 2016 May 1;62(9):385-95. Spanish. PMID 27113062
- [Result] Clua-Espuny JL, Abilleira S, Queralt-Tomas L, Gonzalez-Henares A, Gil-Guillen V, Muria-Subirats E, Ballesta-Ors J. Long-Term Survival After Stroke According to Reperfusion Therapy, Cardiovascular Therapy and Gender. Cardiol Res. 2019 Apr;10(2):89-97. doi: 10.14740/cr839. Epub 2019 Apr 11. PMID 31019638
- [Result] Clua-Espuny JL, Pinol-Moreso JL, Gil-Guillen FV, Orozco-Beltran D, Panisello-Tafalla A, Lucas-Noll J. [The stroke care system in Terres de l'Ebre, Spain, after the implementation of the Stroke Code model: Ebrictus Study]. Med Clin (Barc). 2012 May 19;138(14):609-11. doi: 10.1016/j.medcli.2011.10.004. Epub 2011 Dec 6. Spanish. PMID 22153783